CLINICAL TRIAL: NCT02938026
Title: Changes of Diet, Physical Activity and Sleep Pattern and Their Effects on Glycemic and Weight Control in Hong Kong Chinese Obese Patients With Type 2 Diabetes After Bariatric Surgery Compared to Telephone Intensive Lifestyle Counselling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lorena Tsui Fun Cheung, PhD student in medical science, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lifestyle-002
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus Type 2 in Obese
MeSH Terms: interventions — Bariatric Surgery

ARMS (3):
- Control (No Intervention): Usual care
- Telephone intensive lifestyle counseling (Experimental): Telephone intensive lifestyle counseling
  Interventions: Behavioral: Telephone Intensive Lifestyle Counselling
- Bariatric surgery (Experimental): Bariatric surgery
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery
  Arms: Bariatric surgery
Behavioral: Telephone Intensive Lifestyle Counselling
  Arms: Telephone intensive lifestyle counseling

SUMMARY:
Nutrition therapy is recognized as one of the crucial components for the standard treatment of diabetes along with physical activity and drug therapy. Of note, dietary habits are culture specific and hence understanding the dietary intake, eating behavior and physical activity level of the local population is important to formulate effective nutrition and lifestyle strategies. Weight control is a major therapeutic challenge because many conventionally used anti-diabetic agents, such as sulphonylurea and insulin, can cause weight gain, thus setting up a vicious cycle with increasing insulin resistance due to increasing levels of free fatty acids from adipose tissues . Although intensive face-to-face lifestyle intervention program has showed that even modest weight loss in people with Type 2 diabetes (T2DM) who were overweight or obese was associated with improvements in glycemic control and associated conditions, it may not be feasible in public hospital setting in Hong Kong due to factors such as limited resources, scheduling, patient's employment and willingness for frequent travel to the clinic. Hence, alternative strategies such as a combination of face- to-face individual dietary and lifestyle consultation together with telephone intensive lifestyle reinforcement program will likely to be an useful strategy to engage those obese T2DM patients through frequent individual contacts. On the other hand, bariatric surgery has emerged as an impressive therapeutic option for poorly control obese T2DM patients.

Realizing there is a knowledge gap in understanding the lifestyle factors in the Hong Kong Chinese obese T2DM patients, we therefore propose to conduct a 1-year prospective clinical trial with two main objectives:

1. To study and compare the glycemic and weight improvement after bariatric surgery versus a telephone intensive lifestyle intervention program for 1 year in Hong Kong Chinese obese patients with type 2 diabetes.
2. To investigate the effect of lifestyle factors including dietary intake, eating behaviors and physical activity level on the glycemic and weight control of Hong Kong Chinese obese patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 65 years
2. Chinese ethnicity
3. BMI ≥27.5 kg/m2
4. Diagnosis of T2DM
5. No active cardiovascular diseases
6. ASA grade II or below (for the bariatric surgery group)
7. Able to read Chinese and give informed written consent

Exclusion Criteria:

1. Type 1 diabetes mellitus
2. End-stage renal failure requiring dialysis or chronic kidney disease (CKD) stage 4 or above
3. Malignancy diagnosed within 3 years
4. Major psychiatric illness
5. Pregnancy or lactation
6. Significant anaesthetic risk ASA grade III or above (for the bariatric surgery group)
7. Any medical illness or condition as judged by the investigators as ineligible to participate the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change of HbA1c | 1 year
Change of weight | 1 year

IPD SHARING:
Plan to Share IPD: No